CLINICAL TRIAL: NCT05970939
Title: Development, Reliability and Validity of the Telerehabilitation Usability Questionnaire- TrUQ in Neurological Diseases
Brief Title: Development, Reliability and Validity of the Telerehabilitation Usability Questionnaire- TrUQ
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, principal investigator, Ordu University
Other Study IDs: ND-Development-TrUQ
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Neurological Disease
Keywords: Multiple Sclerosis; Parkinson Disease; Stroke; Usability; Telerehabilitation
MeSH Terms: conditions — Nervous System Diseases; Multiple Sclerosis; Parkinson Disease; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Telerehabilitation Usability: Telerehabilitation Usability Group
  Interventions: Other: Development of the Telerehabilitation Usability Questionnaire

INTERVENTIONS:
Other: Development of the Telerehabilitation Usability Questionnaire — This study will be examined the development, validity, and reliability of the Telerehabilitation Usability Questionnaire in patients with MS.

SUMMARY:
Neurological diseases are central nervous system diseases that cause an increase in the level of disability and limitations in daily life. Multiple Sclerosis (MS), stroke, and Parkinson's Disease (PD) are among the most common apparent neurological diseases, and epidemiological studies show that their prevalence has increased over time worldwide. Although MS, stroke, and PD have different causes and neurological aspects, they generally cause motor, sensory, and/or cognitive impairments, leading to restriction of the individual's activities and participation. Today, physiotherapy and rehabilitation approaches together with optimal medical and surgical treatment are the cornerstones of treatment for these diseases. Recently, it has been stated that various telerehabilitation interventions in the field of physiotherapy and rehabilitation may be an additional option to the rehabilitation approaches applied in the clinic. On the other hand, It is important to evaluate the level of usability in expanding the usability of telerehabilitation services and determining the best telerehabilitation service. For this reason, there is a need for questionnaires investigating the satisfaction level of physiotherapy and rehabilitation applied through telerehabilitation.

DETAILED DESCRIPTION:
Questionnaire items will be created in two stages. First, 5 experts will independently review the literature on "telerehabilitation" and "usability". In addition, these experts will be asked to create a pool of questions based on their experiences in telerehabilitation and by taking the opinions of patients receiving telerehabilitation about usability. Then, 5 experts will come together and obtain a single question pool containing the questions they deem important in their question pool. The second step will involve scaling the elements. In this study, scale items will be scored on a five-point Likert scale, ranging from 1, strongly disagree to 5, strongly agree. Then, it will be applied to a pilot group of 10 people and it will be evaluated whether the items prepared by the experts are understood by the patients. In line with the expert opinion and the result of the pilot study, the final version of the scale will be decided and applied to MS, PD, and stroke patients who make up the study group. Finally, the validity and reliability of the questionnaire will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in research to accept
* Mini-Mental Test score more than or equal 24
* Previously receiving physical therapy through telerehabilitation

Exclusion Criteria:

* Any visual, hearing, and perception problems that may affect the answering the questionnaire items

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurological patients receiving physiotherapy and rehabilitation via telerehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Telerehabilitation Usability Questionnaire in patients with Neurological disease | Baseline
  Patients get a minimum of 0 points (best condition) and a maximum of 4 points (worst condition) for each question on this scale
Telerehabilitation Usability Questionnaire in patients with Neurological disease-Second | he second assessment will be conducted after the one week
  Patients get a minimum of 0 points (best condition) and a maximum of 4 points (worst condition) for each question on this scale

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parmanto B, Lewis AN Jr, Graham KM, Bertolet MH. Development of the Telehealth Usability Questionnaire (TUQ). Int J Telerehabil. 2016 Jul 1;8(1):3-10. doi: 10.5195/ijt.2016.6196. eCollection 2016 Spring. PMID 27563386
- See also: Reference 1 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4985278/